CLINICAL TRIAL: NCT01011010
Title: Phase Ib Clinical Trial of Sorafenib in Combination With Transarterial Chemoembolization (TACE) in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: Sorafenib Tosylate and Chemoembolization With Doxorubicin Hydrochloride and Mitomycin in Treating Patients With Liver Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0902; P30CA016086 (NIH); CDR0000648296 (Other: PDQ number)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Doxorubicin; Mitomycin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): Single Arm Trial
  Interventions: Drug: doxorubicin hydrochloride; Drug: mitomycin C; Drug: sorafenib tosylate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: doxorubicin hydrochloride — TACE (day 18-20): Doxorubicin 50mg and mitomycin C 10mg mixed with lipoidal and injected in proportion to liver volume being treated, followed by embospheres. Administered until there is a "pruned tree" appearance on angiography. If a second TACE is to be performed it should be performed within 8 weeks of the first procedure.
Drug: mitomycin C — TACE (day 18-20): Doxorubicin 50mg and mitomycin C 10mg mixed with lipoidal and injected in proportion to liver volume being treated, followed by embospheres. Administered until there is a "pruned tree" appearance on angiography. If a second TACE is to be performed it should be performed within 8 weeks of the first procedure.
Drug: sorafenib tosylate — Sorafenib 400mg BID continuously post TACE beginning when LFTs return to entry criterion. Discontinue at time of disease progression (progression in a lobe that has already been embolized, new lesions in an untreated lobe, or evidence of extrahepatic progression).
Other: laboratory biomarker analysis — Serum VEGF levels are required: pre TACE (day of procedure, time B), 24 hours post TACE (+/- 6 hours, time C), day 7 post first TACE (± 1 day, time D), day 28 post reinitiation of sorafenib (± 3 days, time E). These levels will not be repeated for patients receiving a second TACE procedure.
Other: pharmacological study — Treatment with sorafenib will continue on a daily basis until disease progression (see definition protocol Section 7) or unacceptable toxicity is encountered. At the end of treatment, no further therapies are currently recommended.

SUMMARY:
RATIONALE: Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as doxorubicin hydrochloride and mitomycin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemoembolization kills tumor cells by carrying drugs directly into the tumor and blocking the blood flow to the tumor. Giving sorafenib tosylate together with chemoembolization may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of sorafenib tosylate when given together with chemoembolization with doxorubicin hydrochloride and mitomycin in treating patients with liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety of sorafenib tosylate when given in combination with transarterial chemoembolization (TACE) comprising doxorubicin hydrochloride and mitomycin C in patients with unresectable hepatocellular carcinoma.

Secondary

* To estimate the time to progression (TTP) in patients treated with this regimen.
* To estimate the overall survival (OS) of patients treated with this regimen.
* To explore correlative relationships between measures of serum VEGF in the peri-procedure TACE period and changes with TACE and sorafenib tosylate as well as patient outcomes (TTP and OS).

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib tosylate twice daily on days 1-14. Patients then undergo transarterial chemoembolization (TACE) comprising doxorubicin hydrochloride and mitomycin C on days 17-19*. Patients then receive oral sorafenib tosylate twice daily beginning after recovery from TACE and continuing in the absence of disease progression or unacceptable toxicity.

NOTE: *A second course of TACE may be administered within 8 weeks after the first TACE procedure.

Blood samples may be collected periodically for biomarker and pharmacokinetic analysis.

After completion of study treatment, patients are followed up at 3-4 weeks and then every 3 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma (HCC), as defined by 1 of the following:

  * Tissue histology

    * Recurrence of previously resected HCC does not require tissue confirmation if there is clear radiographic recurrence, in the judgment of the investigator
  * AFP > 400 ng/mL with compatible mass on MRI
* Locally advanced disease
* Not eligible for surgical resection or immediate liver transplantation OR have refused such procedures
* All disease must be amenable to embolization in one or two procedures
* Measurable disease, according to modified HCC RECIST criteria

  * Must have radiographically documented measurable disease with at least one site of disease that is unidimensionally measurable as ≥ 10 mm on MRI
  * Lesions previously treated by radiofrequency ablation should not represent the only site of measurable disease
* Childs-Pugh score ≤ 7
* No complete thrombosis of the main portal vein

  * If unilateral portal vein thrombosis is present, must demonstrate radiographic evidence of adequate flow to the lobe to be embolized
* No evidence of extrahepatic/metastatic disease, such as lymph node metastases, lung or bone metastases, or peritoneal carcinomatosis

  * Evidence of cirrhosis is acceptable as long as the lab parameters are met
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 9.0 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance ≥ 50 mL/min
* Total bilirubin ≤ 3 mg/dL
* ALT and AST ≤ 5 times ULN
* INR < 1.5
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No other cancer within the past 3 years except for cervical carcinoma in situ, previously treated basal cell carcinoma, or superficial bladder tumors (Ta, Tis, or T1)
* No NYHA class III or IV congestive heart failure
* No unstable angina (anginal symptoms at rest) or new-onset angina within the past 3 months
* No myocardial infarction within the past 6 months
* No cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension (i.e., systolic BP > 150 mm Hg or diastolic BP > 90 mm Hg, despite optimal medical management)
* No venous thrombotic or arterial embolic events (e.g., cerebrovascular accident, including transient ischemic attacks or venous thromboembolism) within the past 6 months
* No pulmonary hemorrhage/bleeding event > CTCAE grade 2 within the past 12 weeks
* No other hemorrhage/bleeding event > CTCAE grade 3 within the past 12 weeks
* No variceal bleeding within past 12 weeks
* No known grade 2 or 3 esophageal varices (endoscopic evaluation is not required for study entry)
* No evidence or history of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 12 weeks
* No serious non-healing wound, ulcer, or bone fracture
* No significant proteinuria (i.e., proteinuria > 1+ on urine dipstick)
* No HIV positivity (by patient report)
* No active hepatitis B or C, unless patient has been on stable medications for ≥ 2 months
* No active clinically serious infections (> grade 2)
* No active gastrointestinal malabsorption problem
* No condition that would impair the patient's ability to swallow whole pills
* No active drug or alcohol abuse
* No known severe hypersensitivity or suspected allergy to sorafenib tosylate, any of its excipients, or other drugs used in this study
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* No prior systemic therapy, embolic therapy, or radiotherapy for HCC (e.g., chemotherapy, transarterial chemoembolization, transarterial embolization, or 90Y microspheres)
* At least 4 weeks since prior liver resection or ablative therapy and recovered
* No prior Raf/MEK/ERK-targeted therapy or VEGF-targeted therapy
* More than 4 weeks since prior participation in any investigational drug study
* More than 12 weeks since prior major surgery or open biopsy

  * Prior core liver biopsy allowed
* No concurrent antiretroviral therapy for HIV
* No concurrent chronic anticoagulation (other than 1 mg of warfarin daily for port patency)
* No concurrent St. John wort or rifampin
* No other concurrent anticancer therapy, radiotherapy, or investigational therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07-22 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity as assessed by NCI CTCAE v3.0 criteria | 3 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Correlative studies | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hanna H. Sanoff, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/results?cond=&term=NCT01011010&cntry=&state=&city=&dist=